CLINICAL TRIAL: NCT06796322
Title: A Prospective, Multicenter, Non-randomized, Open-label, Self-controlled, Paired Clinical Trial to Evaluate the Effectiveness and Safety of a Non-invasive Blood Glucose Meter Compared With Laboratory Detection in Diabetic Patients
Brief Title: Clinical Evaluation of Non-invasive Blood Glucose Meter
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai 10th People's Hospital (Other); Hanchuan People's Hospital (Unknown)
Responsible Party: Principal Investigator, Wang Weiqing, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: JGKJ01202401
Record Dates: First submitted 2025-01-13; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Glucose detection
Masking Description: Masking Description
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-invasive blood glucose meter (Experimental): Non-invasive blood glucose meter by the non-invasive blood glucose meter using a Raman spectrum measurement system.
  Interventions: Device: non-invasive blood glucose meter
- Fully automatic laboratory biochemical analyzer (Other): Fully automatic laboratory biochemical analyzer (the primary control group) using the hexokinase method to measure venous plasma blood glucose.
  Interventions: Device: fully automatic laboratory biochemical analyzer
- Fingertip capillary blood sample (Other): Fingertip capillary blood sample (the secondary control group) to detect fingertip capillary blood glucose.
  Interventions: Device: fingertip capillary blood glucose meter

INTERVENTIONS:
Device: non-invasive blood glucose meter — Blood glucose were detected by non-invasive glucose meter at four time points, namely fasting, 1 hour post breakfast, 2 hours post breakfast, and 3 hours post breakfast.
  Arms: Non-invasive blood glucose meter
Device: fully automatic laboratory biochemical analyzer — Blood glucose were detected by fully automatic laboratory biochemical analyzer using plasma sample at four time points, namely fasting, 1 hour post breakfast, 2 hours post breakfast, and 3 hours post breakfast.
  Arms: Fully automatic laboratory biochemical analyzer
Device: fingertip capillary blood glucose meter — Blood glucose were detected by fingertip capillary blood sample at four time points, namely fasting, 1 hour post breakfast, 2 hours post breakfast, and 3 hours post breakfast.
  Arms: Fingertip capillary blood sample

SUMMARY:
This trial is a prospective, multicenter, non-randomized, open-label, self-controlled, paired design clinical study, which will be conducted in 3 research centers, with a total of 210 subjects enrolled, including diabetic patients aged 18 years and above and some healthy subjects. After screening, each eligible subject will have their blood glucose measured simultaneously at specified time points using three methods: non-invasive blood glucose meter (the experimental group), fully automatic laboratory biochemical analyzer (the primary control group) using the hexokinase method to measure venous plasma blood glucose, and fingertip capillary blood sample (the secondary control group) to detect fingertip capillary blood glucose. The aim of this trial is to evaluate the efficacy and safety of the non-invasive blood glucose meter for blood glucose measurement in diabetic patients.

DETAILED DESCRIPTION:
After screening, the qualified subjects complete the blood glucose measurement in three ways at the following time points on the test day, namely, fasting blood glucose before breakfast, 1 hour post breakfast, 2 hours post breakfast, and 3 hours post breakfast.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for healthy subjects:

* Male or female, aged >=18 years.
* Fully understand the nature, significance, possible benefits, possible inconveniences or potential risks of this research, and should also understand the research procedures, be willing to complete the entire research process, and provide written consent form.

Inclusion Criteria for patients with type 2 diabetes:

* Male or female, aged >=18 years.
* Previously diagnosed type 2 diabetes according to WHO criteria of 1999.
* Fully understand the nature, significance, possible benefits, possible inconveniences or potential risks of this research, and should also understand the research procedures, be willing to complete the entire research process, and provide written consent form.

Exclusion Criteria:

Exclusion Criteria for healthy subjects:

* There are injuries, scars, obvious pigmentation and other factors that interfere with the detection of the palm skin to be tested.
* Allergy to lasers.
* Had diabetes history or fasting blood glucose (FPG) >= 6.1 mmol/L or glycated hemoglobin (HbA1c) >= 5.7% during the screening period.
* Alcohol dependency or drug abuse.
* Those who have participated in clinical trials of other drugs within 3 months before screening (since the last visit of the previous trial).
* Pregnancy or lactation period.
* Difficulty in venous blood collection or fainting of needles or blood.
* Other circumstances that the investigator considers inappropriate to participate in the study.

Exclusion Criteria for patients with type 2 diabetes:

* There are injuries, scars, obvious pigmentation and other factors that interfere with the detection of the palm skin to be tested.
* Allergy to lasers.
* Type 1 diabetes, monogenic mutant diabetes, pancreatic damage, or secondary diabetes of other causes should be excluded.
* Severe structural heart disease, such as congenital heart disease, rheumatic heart disease, hypertrophic or dilated cardiomyopathy, chronic congestive heart failure (NYHA≥III); acute myocardial infarction within 12 months before enrollment; history of severe liver or kidney dysfunction (eGFR < 60 ml/min/1.73m2 calculated by MDRD formula at screening period); and mental disorders, etc.
* With a history of acute complications of diabetes within 3 months before enrollment; or severe diabetes-related complications.
* Alcohol dependency or drug abuse.
* Those who have participated in clinical trials of other drugs within 3 months before screening (since the last visit of the previous trial).
* Pregnancy or lactation period.
* Difficulty in venous blood collection or fainting of needles or blood.
* Other circumstances that the investigator considers inappropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Consensus Error Grid (CEG) for venous plasma glucose and glucose values measured by non-invasive glucose meter of mμSORS at each time point indicated. | 3 months
  Glucose will be measured using both intravenous sampling (plasma) and non-invasive meter of mμSORS synchronously.

SECONDARY OUTCOMES:
The MARD were evaluated for non-invasive glucose meter using venous plasma glucose as the control. | 3 months
  The interval between the two methods is less than 10 minutes at each point.
The ±20% agreement were evaluated for non-invasive glucose meter using venous plasma glucose as the control. | 3 months
  The interval between the two methods is less than 10 minutes at each point.
The point proportion of A+B region of Clarke error grid analysis were evaluated for non-invasive glucose meter using venous plasma glucose as the control. | 3 months
  The interval between the two methods is less than 10 minutes at each point.
The regression analysis were evaluated for non-invasive glucose meter using venous plasma glucose as the control. | 3 months
  The interval between the two methods is less than 10 minutes at each point.
The bland-Altman analysis were evaluated for non-invasive glucose meter using venous plasma glucose as the control. | 3 months
  The interval between the two methods is less than 10 minutes at each point.
The MARD were evaluated for non-invasive glucose meter using fingertip capillary blood sample as the control. | 3 months
  The interval between the two methods is less than 10 minutes at each point.
The ±20% agreement were evaluated for non-invasive glucose meter using fingertip capillary blood sample as the control. | 3 months
  The interval between the two methods is less than 10 minutes at each point.
The point proportion of A+B region of Clarke error grid analysis were evaluated for non-invasive glucose meter using fingertip capillary blood sample as the control. | 3 months
  The interval between the two methods is less than 10 minutes at each point.
The regression analysis were evaluated for non-invasive glucose meter using fingertip capillary blood sample as the control. | 3 months
  The interval between the two methods is less than 10 minutes at each point.
The bland-Altman analysis were evaluated for non-invasive glucose meter using fingertip capillary blood sample as the control. | 3 months
  The interval between the two methods is less than 10 minutes at each point.
Incidence of Treatment-Emergent Adverse Events | 3 months
  Safety in the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Weiqing Wang, Dr., Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China